CLINICAL TRIAL: NCT02662920
Title: Investigating the Prevalence and Prognostic Importance of Polypharmacy in Adults Treated for Newly Diagnosed Acute Myelogenous Leukemia (AML)
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00014134; CCCWFU 22410 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: ACUTE MYELOGENOUS LEUKEMIA
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention

SUMMARY:
Prevalence and prognostic significance of polypharmacy has not been evaluated in adults undergoing treatment for AML. Investigating the significance of polypharmacy in this population may help improve patient assessment and provide an opportunity to design simple interventions to minimize unnecessary morbidity associated with treatment.

DETAILED DESCRIPTION:
The incidence of acute myelogenous leukemia (AML) increases with age. Older AML patients, generally defined by age 60 years and above, have worse treatment outcomes than younger patients. While selected older patients can benefit from standard therapies, as a group they experience increased treatment-related toxicity, decreased remission rates, decreased disease-free survival and decreased overall survival. Outcome disparity is in part explained by age related biologic features. Older patients are more likely to present with unfavorable cytogenetic abnormalities, multidrug resistance phenotypes, and secondary AML. However, even older adults with favorable tumor biology have a worse prognosis compared to younger patients. Patient-specific factors including impaired physical function and comorbidity independently predict increased treatment toxicity and decreased survival. Improving patient assessment strategies is critical to identify those patients who are most likely to benefit from induction and post-remission therapies.

Treatment decision-making for older adults is hampered by the difficulty of accurately predicting vulnerability to toxicity. Increasing age alone is a risk factor for poor response to therapy. Older adults of the same chronologic age represent a heterogeneous population. Multiple patient-specific factors may impact an older adult's ability to tolerate tumor burden and treatments. Comorbid disease, functional status and cognitive status are examples of factors that reflect an individual patient's reserve capacity; none of these can be adequately assessed with chronologic age alone.

Translating geriatric assessment strategies into the evaluation of older patients with acute leukemia should help refine the treatment approach to this population. One strategy commonly used in geriatric medicine is the comprehensive geriatric assessment (CGA). CGA refers to a multidisciplinary evaluation of geriatric domains, including comorbid disease, physical function, cognitive function, psychological state, nutritional status, and medication management. In older cancer patients CGA can identify problems that may interfere with cancer treatment and is recommended by the NCCN Guidelines for "Senior Adult Oncology". The optimal measures to use and how to change management based on results are less clear.

Medication management may be of particular importance for older adults with AML due to the potentially high prevalence of polypharmacy in this population. Studies of older adults with cancer report average numbers of medications ranging from 4-9. These numbers may be higher for patients being actively treated for acute leukemia. Polypharmacy is associated with increased adverse drug reactions and increased risk of drug-drug interactions. Careful medication review with discontinuation of potentially unnecessary or inappropriate medications may minimize negative consequences of polypharmacy.

To date, however, prevalence and prognostic significance of polypharmacy has not been evaluated in adults undergoing treatment for AML. Investigating the significance of polypharmacy in this population may help improve patient assessment and provide an opportunity to design simple interventions to minimize unnecessary morbidity associated with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized between January 2004 and December 2009 with newly diagnosed AML
* Age ≥60 years at the time of diagnosis
* Received treatment while hospitalized for AML

Exclusion Criteria:

* 30-day mortality data unavailable

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age ≥60 who received treatment while hospitalized for AML
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of polypharmacy in adults ≥60 years of age hospitalized for treatment of newly diagnosed AML | Day 1 (admission)
  Number of medications at baseline
Prevalence of polypharmacy in adults ≥60 years of age hospitalized for treatment of newly diagnosed AML | Through hospitilization, an average of 30 days
  Number of medications at discharge